CLINICAL TRIAL: NCT05280509
Title: An Open-Label, Multicenter, Phase 1b/2 Study of the Safety and Efficacy of TL-895 Combined With Ruxolitinib in Janus-associated Kinase Inhibitor (JAKi) Treatment-Naïve Myelofibrosis (MF) Subjects and Subjects With MF Who Have a Suboptimal Response to Ruxolitinib
Brief Title: Study of TL-895 Combined With Ruxolitinib in JAKi Treatment-Naïve MF Subjects and Subjects With MF Who Have a Suboptimal Response to Ruxolitinib
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Telios Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TL-895-209
Record Dates: First submitted 2022-03-05; First posted 2022-03-15 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Myelofibrosis; Primary Myelofibrosis; Post-PV MF; Post-ET Myelofibrosis
Keywords: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Intervention Model Description: Phase 1b - Dose Escalation Design Phase 2 - Dose Expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1b - Dose Level 1 (Experimental): 150 mg of TL-895 will be administered orally, twice daily (BID) continuously starting on Day 1 in a 28-day cycle combined with the subject's pre-study stable dose of ruxolitinib.
  Interventions: Drug: TL-895; Drug: Ruxolitinib
- Phase 1b - Dose Level 2 (Experimental): 300 mg of TL-895 will be administered orally, twice daily (BID) continuously starting on Day 1 in a 28-day cycle combined with the subject's pre-study stable dose of ruxolitinib.
  Interventions: Drug: TL-895; Drug: Ruxolitinib
- Phase 1b - Dose Level 3 (Experimental): 450 mg of TL-895 will be administered orally, twice daily (BID) continuously starting on Day 1 in a 28-day cycle combined with the subject's pre-study stable dose of ruxolitinib.
  Interventions: Drug: TL-895; Drug: Ruxolitinib
- Phase 2 - Cohort 1 JAKi treatment-naïve MF (Experimental): The RP2D of TL-895 as determined in Phase 1b will be administered orally, twice daily (BID) continuously starting on Day 1 in a 28-day cycle.
  The dose of ruxolitinib will be based on the subject's baseline platelet count.
  Interventions: Drug: TL-895; Drug: Ruxolitinib
- Phase 2 - Cohort 2 suboptimal response to Ruxolitinib (Experimental): The RP2D of TL-895 as determined in Phase 1b will be administered orally, twice daily (BID) continuously starting on Day 1 in a 28-day cycle.
  The dose schedule will be the stable ruxolitinib dose schedule as the subject is currently taking prior to entry into the study.
  Interventions: Drug: TL-895; Drug: Ruxolitinib

INTERVENTIONS:
Drug: TL-895 — TL-895 is an experimental tyrosine kinase inhibitor anticancer drug taken by mouth.
Drug: Ruxolitinib — Ruxolitinib is an FDA-approved janus kinase inhibitor anticancer drug taken by mouth.
  Other Names: Jakafi; Jakavi

SUMMARY:
This study evaluates TL-895, a potent, orally-available and highly selective irreversible tyrosine kinase inhibitor for the treatment of Myelofibrosis. Participants must have MF (PMF, Post PV MF, or Post ET MF) who are JAKi treatment-naïve or those who have a suboptimal response to ruxolitinib.

ELIGIBILITY:
Inclusion Criteria:

Subjects with suboptimal response to ruxolitinib:

* Treatment with at a stable dose of ruxolitinib prior to study entry
* Subjects ≥ 18 years of age and able to provide informed consent.
* Confirmed diagnosis of PMF, post-PV MF, or post-ET MF, as assessed by treating physician according to the World Health Organization (WHO) criteria
* High-risk, intermediate-2 risk, or intermediate-1 risk, defined by Dynamic International Prognostic System (DIPSS)
* Palpable spleen measuring ≥ 5 cm below the left lower coastal margin (LLCM) or spleen volume of ≥ 450 cm3 by MRI or CT scan assessment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Adequate hematological, hepatic, & renal function.

Exclusion Criteria:

Treatment-naive subjects:

* Prior treatment with any JAKi

Subjects with suboptimal response to ruxolitinib:

* Documented disease progression while on ruxolitinib treatment

All subjects:

* Prior splenectomy or splenic irradiation within 24 weeks prior to first dose of study treatment
* Prior treatment with a BTK or BMX inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Phase 1b - Recommended Phase 2 dose of TL-895 in combination with ruxolitinib | 28 days
  Dose-limiting toxicities (DLTs) will be used to establish the maximum-tolerated dose (MTD) of TL-895 in combination with ruxolitinib. The safety review committee (SRC) will determine the RP2D based on safety and efficacy data of the combination of TL-895 and ruxolitinib.
Phase 2 - Spleen Volume Reduction (SVR) at Week 24 | 24 Weeks
  The proportion of subjects achieving SVR of ≥35% at Week 24 by magnetic resonance imaging (MRI) or computed tomography (CT) scan.

SECONDARY OUTCOMES:
Phase 1b - Spleen Volume Reduction (SVR) at Week 24 | 24 Weeks
  The proportion of subjects achieving ≥35% SVR at Week 24 by MRI or CT scan.
Phase 1b - TSS reduction at Week 24 | 24 Weeks
  The proportion of subjects achieving ≥50% reduction in TSS at Week 24 by Myelofibrosis Symptom Assessment Form (MFSAF) v4.0.
Phase 2 - TSS reduction at Week 24 | 24 Weeks
  The proportion of subjects achieving ≥50% reduction in TSS at Week 24 by MFSAF v4.0.
DOR Spleen | 48 Months
  Time from initial SVR of ≥ 35% by MRI/CT until the first occurrence of disease progression or death
Progression Free Survival | 48 Month
  Time from first dose to progression or death from any cause.
Overall Survival | 48 Months
  Time from first dose to death from any cause

CONTACTS AND LOCATIONS:
Locations (19):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Gabrail Cancer Center, Canton, Ohio
  - University of Cincinnati (UC), Cincinnati, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- France (5):
  - CHU Angers, Angers
  - AP-HM - Hôpital de la Timone, Marseille
  - CHU de Nice - Hopital L'Archet II, Nice
  - Hôpital Saint Louis - AP-HP, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- Germany (2):
  - Marien Hospital Duesseldorf, Düsseldorf
  - Klinik fur Innere Medizin IV - Hamatologie/Onkologie, Universitatsklinikum Hall, Halle
- Italy (3):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - Policlinico di Sant'Orsola, Bologna
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan
  - Azienda Ospedaliera di Perugia-Ospedale S. Maria della Misericordia, Perugia
- Pratia Onkologia Katowice, Katowice, Poland
- Spain (4):
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Quironsalud de Zaragoza, Zaragoza